CLINICAL TRIAL: NCT02433405
Title: Serum Amyloid A Protein And Fetuin A Protein Levels In Periodontal Health And Disease
Brief Title: Serum Amyloid A Protein And Fetuin A Levels
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ÇİĞDEM COŞKUN TÜRER, Dr., Bulent Ecevit University
Other Study IDs: SAAFA1
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Periodontal Diseases
Keywords: Serum Amyloid A; Fetuin-A; gingival crevicular fluid; serum; periodontal diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — alpha-2-HS-Glycoprotein; Serum Amyloid A Protein

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid and Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Chronic Periodontitis-serum amyloid A, Fetuin-A
  Interventions: Biological: Fetuin-A; Biological: Serum Amyloid A
- Group 2: Plaque induced Gingivitis-serum amyloid A, Fetuin-A
  Interventions: Biological: Fetuin-A; Biological: Serum Amyloid A
- Group 3: Control Group-serum amyloid A, Fetuin-A
  Interventions: Biological: Fetuin-A; Biological: Serum Amyloid A

INTERVENTIONS:
Biological: Fetuin-A — Acute phase protein
Biological: Serum Amyloid A — Acute phase protein

SUMMARY:
The purpose of this study was to evaluate acute phase proteins (APPs) Fetuin-A and Serum Amyloid A (SAA) levels in gingival crevicular fluid (GCF) and serum samples in periodontal health and disease.

DETAILED DESCRIPTION:
The study population consisted totally 60 subjects consulted to Bulent Ecevit University, Faculty of Dentistry, Department of Periodontology whose age and sex were matched.

According to study design, subjects were divided into three groups based on their periodontal parameters. Patients suffering from chronic periodontitis formed the group 1 (n: 20), patients with plaque induced gingivitis formed the group 2 (n:20) and periodontal healthy patients were inserted in group 3 (n:20).

After gently drying the area, GCF was sampled with filter paper using the intracrevicular method (Periopaper, ProFlow, Inc., Amityville, New York, USA).Two milliliters (ml) of peripheral blood was collected from each individual with sterile syringe from the antecubital fossa by venipuncture, and to separate serum component sample centrifuged at 3000g for 5 min, and immediately stored at -40°C until assayed.

The quantity of Fetuin-A and SAA protein concentration in the samples were analyzed by sandwich enzyme-linked immunosorbent assay (ELISA) procedures using commercially available kits.

The Spearman's rank correlation test was used to detect the relationship between GCF and serum SAA and Fetuin-A with GI and CAL. All tests were performed using statistical software (SPSS Inc., version 22.0, Chicago, IL, USA). The mean ± standard deviation with mean rank values were calculated for each parameter, based on the patients as the statistical unit. P < 0.05 was considered to be statistically significant.

ELIGIBILITY:
Group 1 Inclusion Criteria:

* GI>1, PPD≥5mm, CAL≥5mm with alveolar bone loss radiographically.
* Systematically healthy patients

Group 2 Inclusion Criteria:

* No alveolar bone and attachment loss
* Inflammation signs such as redness, edema and increased BOP levels,
* GI≥2, PPD≤3mm, CAL≤3mm.
* Systematically healthy patients

Group 3 Inclusion Criteria:

* No bone and attachment loss,
* GI=0, PPD≤3mm, CAL≤3mm
* Systematically healthy patients

Exclusion Criteria for all groups:

* Aggressive Periodontitis,
* Oral pathologies,
* Patients with any other systemic diseases,
* Pregnant women and those in the lactation period,
* Patients with smoking habit and taking medication
* Patients received periodontal therapy in last 6 months

Ages: 28 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted totally 60 subjects whose age (28-45) and sex (33 men, 27 female) were matched.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Serum Amyloid A (SAA) levels as an inflammatory marker in periodontal disease both in serum and GCF | Day 0

SECONDARY OUTCOMES:
Fetuin-A levels as an inflammatory marker in periodontal disease both in serum and GCF | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: ÇİĞDEM COŞKUN TÜRER, PhD, Principal Investigator — BULENT ECEVIT UNIVERSITY FACULTY OF DENTISTRY DEPARTMENT OF PERIODONTOLOGY